CLINICAL TRIAL: NCT06244186
Title: The Effect of Lactobacillus Delbrueckii Subsp. Bulgaricus on Human's Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: CMUH110-REC2-070
Record Dates: First submitted 2024-01-02; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
Keywords: Lactobacillus delbrueckii subsp. Bulgaricus; weight reduction; health care
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the placebo or probiotics group, receiving continuous administration for 12 weeks. Measurements of weight, BMI, and body fat were taken on days 0, 28, 56, and 84 of the treatment period. Additionally, 15 mL of fasting blood was drawn on both the first and 84th day.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Take one packet (6 grams) of powder orally once daily. The probiotics contain fruit juice powder (strawberry, cranberry, black currant), sucralose, anhydrous citric acid, maltodextrin, silicon dioxide, and Lactobacillus delbrueckii subsp. Bulgaricus.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo contains fruit juice powder (strawberry, cranberry, black currant), sucralose, anhydrous citric acid, maltodextrin, and silicon dioxide.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics contains a probiotic known as Lactobacillus delbrueckii subsp. Bulgaricus, a key bacterium utilized in the production of yogurt, cheeses, and various naturally fermented products. Studies suggest that the metabolites of Lactobacillus bulgaricus can enhance immunity and digestion, reduce the risk of infection, and lower blood cholesterol levels. The composition of probiotics has been developed by TCI CO., Ltd.
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo is provided by TCI CO., Ltd.
  Arms: Placebo

SUMMARY:
To evaluate the improvement in weight, body fat, and BMI after adding probiotics as a once-daily therapy for 84 days in overweight individuals.

DETAILED DESCRIPTION:
The study product contains Lactobacillus delbrueckii subsp. Bulgaricus at a concentration of 1x10^8 CFU in each 100 mg. The objective of this study is to evaluate the benefits of probiotics as an add-on therapy in overweight individuals by assessing the improvements in weight, body fat, and BMI after adding probiotics as a once-daily therapy for 84 days.

A randomized, two-regimen, placebo-controlled, parallel design is employed in this study, where each subject will receive either probiotics or a placebo. The add-on study product will be administered once daily for 84 days. The benefits will be assessed at baseline and subsequently on study days 28, 56, and 84, focusing on parameters such as weight, body fat, and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Overweight (BMI ≥ 23) or body fat percentage ≥ 25% for males and ≥ 30% for females
* Having any of the following risk factors: Atherosclerotic cardiovascular disease, type 2 diabetes, age ≥ 45 years for males, ≥ 55 years for females or postmenopausal, hypertension, dyslipidemia (total cholesterol > 200 mg/dL or low-density lipoprotein cholesterol > 130 mg/dL or triglycerides > 130 mg/dL), high-density lipoprotein cholesterol < 40 mg/dL
* If routinely taking medication for lowering blood glucose, blood pressure, or lipid levels, there should not be significant dosage changes within the past three months
* Being willing to participate after receiving an explanation from the physician, completing the trial plan, and signing the consent form

Exclusion Criteria:

* History of diabetic ketoacidosis
* Medical records indicating the occurrence of cerebrovascular disease, acute myocardial infarction, coronary artery bypass surgery, placement of coronary artery stents, or peripheral vascular disease within the last 6 months
* Occurrence of acute infectious diseases within the last month and antibiotic use for > 7 days
* Short-term use of steroids, NSAIDs, immunosuppressive drugs, interferons, immunomodulators, or any changes in the dose of long-term medications within the last month
* Use of any weight-loss drugs in the last three months (including Orlistat, Lorcaserin, and liraglutide)
* History of any cancer or undergoing cancer treatment in the past 5 years
* Abnormal liver function (GOT or GPT greater than 3 times the normal upper limit) or liver cirrhosis
* Impaired kidney function (eGFR < 30 mL/min/1.73 m2)
* History of alcohol abuse
* Participation in any other interventional clinical research within the last month
* Pregnant and breastfeeding women
* History of allergy to the investigational product
* Participants deemed unsuitable for inclusion by the principal investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Body weight | 84 days
  Comparing the changes between Day 0 and Day 84
Body fat | 84 days
  Comparing the changes between Day 0 and Day 84
BMI | 84 days
  Comparing the changes between Day 0 and Day 84

SECONDARY OUTCOMES:
ALT and AST (U/L) in Blood composition | 84 days
  Comparing the changes in ALT and AST (alanine aminotransferase, aspartate aminotransferase) in the blood between Day 0 and Day 84
CRE, BUN and GLU-AC (mg/dL) in Blood composition | 84 days
  Comparing the changes in CRE, BUN, and GLU-AC (creatinine, blood urea nitrogen, fasting blood glucose) in the blood between Day 0 and Day 84
Changes in glycated hemoglobin | 84 days
  Comparing the changes in hemoglobin A1c between Day 0 and Day 84.
Changes in CHOL, TG, HDL and LDL-C (mg/dL) in Blood composition | 84 days
  Comparing the changes in CHOL, TG, HDL, and LDL-C (cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) between Day 0 and Day 84.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chin Huang, PhD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT06244186/Prot_SAP_000.pdf